CLINICAL TRIAL: NCT02880397
Title: Clinical And Microbiological Efficacy Of 4% Garcinia Mangostana L.Pericarp Gel As A Local Drug Delivery In The Treatment Of Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Garcinia Mangostana L.Pericarp Gel as a Local Drug Delivery in Treatment of Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Dr. Jaideep Mahendra, Meenakshi Ammal Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAHER - REG 2214001
Record Dates: First submitted 2016-08-11; First posted 2016-08-26 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Generalized Chronic Periodontitis
Keywords: Anti-inflammatory agents, antimicrobials, Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Garcinia Mangostana (Active Comparator): The constituents of mangostana containing gel were prepared under the following proportions: Mangostana powder - 4gm, Gelatin - 12gm, Glycerin (wetting agent) - 0.2ml, Peppermint oil (flavouring agent) - 0.1ml, sodium saccharine (sweetening agent) - 0.1ml and purified water q.s 100ml.
  Interventions: Drug: Garcinia mangostana
- Placebo gel (Placebo Comparator): The placebo gel was prepared with Gelatin - 12gm, Glycerin (wetting agent) - 0.2ml, Peppermint oil (flavouring agent) - 0.1ml, sodium saccharine (sweetening agent) - 0.1ml and purified water q.s 100ml excluding the active ingredient mangostana powder - 4 mg and maintaining same physical properties such as color and taste.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Garcinia mangostana — The properties of mangostana includes antibacterial, antifungal, anti-inflammatory, anti-microbial, antioxidant, anticancer, anti-proliferative, pro-apoptotic, aromatase inhibitory properties
  Other Names: Mangosteen
  Arms: Garcinia Mangostana
Drug: Placebo gel — The properties of placebo includes antibacterial, antifungal, anti-inflammatory, anti-microbial, antioxidant, anticancer, anti-proliferative, pro-apoptotic, aromatase inhibitory properties
  Other Names: Placebo
  Arms: Placebo gel

SUMMARY:
A single-center, randomized controlled clinical trial was done to assess the periodontal status of the individuals and the presence of red complex microorganisms (RCM) such as Treponema denticola, Porphyromonas.gingivalis and Tannerella.forsythia in the subgingival tissues of periodontal pockets at baseline followed by the application of mangostana gel as an adjunct to scaling and root planing. The periodontal parameters and RCM were again assessed at 3rd month and compared with the placebo group.

DETAILED DESCRIPTION:
Background: The study aim to assess the periodontal status of individuals and the presence of red complex microorganisms (RCM) such as Treponema denticola (T.d), Porphyromonas gingivalis (P.g) and Tannerella forsythia (T.f) in the subgingival tissues of periodontitis subjects before and after the application of 4% mangostana gel (MGA) as an adjunct to scaling and root planing.

Methods: 25 sextants (MGA group) were treated with scaling and root planing (SRP) and subgingival application of mangostana gel used as local drug delivery (LDD). 25 sextants (Placebo group) were treated with SRP and placebo gel. Clinical parameters were recorded and the presence of RCM were assessed at baseline and at 3rd month.

Statistical Analysis: The mean probing pocket depth, clinical attachment level, bleeding index, plaque index were assessed at 0th day and 3rd month and compared between the groups using one way analysis of co-variance (ANCOVA). Intra-group comparison (MGA) for the presence of T.d, from baseline to 3rd month and inter-group comparison (MGA & Placebo) at 3rd month was done using Fischer exact test. In both MGA and placebo group, the presence of T.d in subgingival tissues was compared with the clinical parameters at 3rd month using student's t-test. The p ≤ 0.05 was chosen as a level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30 to 65 years
* Systemically healthy subjects with chronic periodontitis

Exclusion Criteria:

* aggressive periodontitis,
* systemic disorders,
* known or suspected allergy to the MGA/placebo group,
* pregnant and lactating females,
* long term steroid medication,
* smokers,
* alcoholics,
* immunocompromised individuals and
* those with history of antibiotic or periodontal therapy in preceding 6 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of 4% mangostana in chronic periodontitis patients from baseline to 3 months. | 3 months
  probing pocket depth was measured using Williams periodontal probe with the measurement of 0 to 9 mm and the criteria is as follows - 2 to 4 mm for gingivitis, 4 to 5 mm for slight periodontitis, 6 to 7 mm for moderate periodontitis and > 7 mm for advanced periodontal disease.
  Clinical attachment level was measured from cemento-enamel junction to the base of the pocket using Williams periodontal probe with the criteria of 1 to 2 mm for slight periodontitis, 3 to 4 mm for moderate periodontits and greater or equal to 5 mm for severe periodontitis.

SECONDARY OUTCOMES:
Microbiological efficacy of 4% mangostana in chronic periodontitis patients from baseline to 3 months. | 3 months
  Red complex microorganisms such as Porphyromonas gingivalis, Tannerella forsythia and Treponema denticola were analysed using 16S rRNA gene amplification by polymerase chain reaction for their absence as '0' and presence as '1'.

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, Principal Investigator — Meenakshi Ammal Dental College and Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steinmetz KA, Potter JD. Vegetables, fruit, and cancer prevention: a review. J Am Diet Assoc. 1996 Oct;96(10):1027-39. doi: 10.1016/S0002-8223(96)00273-8. PMID 8841165
- [Result] Shankaranarayan D, Gopalakrishnan C, Kameswaran L. Pharmacological profile of mangostin and its derivatives. Arch Int Pharmacodyn Ther. 1979 Jun;239(2):257-69. PMID 314790
- [Result] Rassameemasmaung S, Sirikulsathean A, Amornchat C, Maungmingsook P, Rojanapanthu P, Gritsanaphan W. Topical application of Garcinia mangostana L. pericarp gel as an adjunct to periodontal treatment. Complement Ther Med. 2008 Oct;16(5):262-7. doi: 10.1016/j.ctim.2007.12.004. PMID 19186342